CLINICAL TRIAL: NCT00004246
Title: A Phase I Study of Fludarabine With Radiotherapy in Patients With Locally Advanced Squamous Cell Carcinoma of the Head and Neck
Brief Title: Radiation Therapy Plus Fludarabine in Treating Patients With Locally Advanced Cancer of the Mouth, Pharynx, or Larynx
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ID95-038; P30CA016672 (NIH); P01CA006294 (NIH); MDA-ID-95038 (Other: UT MD Anderson Cancer Center); NCI-H99-0046; CDR0000067492 (Registry Identifier: NCI PDQ)
Record Dates: First submitted 2000-01-28; First posted 2004-05-03 (Estimated); Last update posted 2018-10-25 (Actual); Status verified 2018-10

CONDITIONS: Head and Neck Cancer
Keywords: Radiation Therapy; RT; Radiotherapy; Fludarabine; Fludara; Fludarabine Phosphate; stage III squamous cell carcinoma of the lip and oral cavity; stage IV squamous cell carcinoma of the lip and oral cavity; stage III squamous cell carcinoma of the oropharynx; stage IV squamous cell carcinoma of the oropharynx; stage III squamous cell carcinoma of the nasopharynx; stage IV squamous cell carcinoma of the nasopharynx; stage III squamous cell carcinoma of the hypopharynx; stage IV squamous cell carcinoma of the hypopharynx; stage III squamous cell carcinoma of the larynx; stage IV squamous cell carcinoma of the larynx
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — fludarabine phosphate; fludarabine; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- RT + Fludarabine (Experimental): Radiotherapy (RT) on Days 1-5 for 7 weeks + Fludarabine IV, 3-4 hours prior to daily RT, Days 1-5 of weeks 6 and 7 of RT
  Interventions: Drug: Fludarabine Phosphate; Radiation: Radiation Therapy (RT)

INTERVENTIONS:
Drug: Fludarabine Phosphate — IV on days 1-5 of weeks 6 and 7 of radiotherapy, administered 3-4 hours prior to daily radiotherapy.
  Other Names: Fludara; Fludarabine
Radiation: Radiation Therapy (RT) — Days 1-5 for 7 weeks
  Other Names: radiotherapy

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to damage tumor cells. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining chemotherapy with radiation therapy may kill more tumor cells.

PURPOSE: Phase I trial to study the effectiveness of radiation therapy plus fludarabine in treating patients who have locally advanced cancer of the mouth, pharynx, or larynx.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the maximum tolerated dose of fludarabine that can be given during the sixth and seventh weeks of radiotherapy in patients with locally advanced squamous cell carcinoma of the oral cavity, pharynx, or larynx, based on the systemic toxicity of the drug and the acute mucosal reactions in the irradiated fields. II. Document the qualitative and quantitative toxicity of this combination therapy in this patient population.

OUTLINE: This is a dose escalation study of fludarabine. Patients receive radiotherapy on days 1-5 for 7 weeks. Patients receive fludarabine IV on days 1-5 of weeks 6 and 7 of radiotherapy. Fludarabine is administered 3-4 hours prior to daily radiotherapy. Cohorts of 3 patients receive escalating doses of fludarabine until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose that produces a severe toxicity rate nearest to 20%. Patients are followed every 4 weeks after the completion of treatment until acute reactions have resolved, then every 3 months for 2 years, every 4 months for 1 year, and then every 6 months for 2 years.

PROJECTED ACCRUAL: A maximum of 18 patients will be accrued for this study within 1.5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed squamous cell carcinoma of the oral cavity, pharynx, or larynx for which surgery would result in significant functional impairment Stage III or IV (T3-4 or N2-3) No distant metastases

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Zubrod 0-2 Life expectancy: At least 6 months Hematopoietic: Granulocyte count at least 1,500/mm3 Platelet count at least 150,000/mm3 Hepatic: Bilirubin no greater than 1.5 mg/dL SGOT less than 4 times upper limit of normal PT/PTT normal Renal: Creatinine no greater than 1.5 mg/dL Other: Not pregnant or nursing Fertile patients must use effective contraception No other concurrent acute illness or infection

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No prior chemotherapy Endocrine therapy: Not specified Radiotherapy: No prior radiotherapy Surgery: See Disease Characteristics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 1995-06-07 (Actual); Primary Completion 2002-12-02 (Actual); Study Completion 2002-12-02 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of Fludarabine During Sixth & Seventh Weeks of Radiotherapy | Every 4 weeks
  MTD based on systemic toxicity of drug and acute mucosal reactions in the irradiated fields.

CONTACTS AND LOCATIONS:
Overall Officials: K. Kian Ang, MD, PhD, Study Chair — M.D. Anderson Cancer Center
Locations (1):
- University of Texas - MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center Website — http://www.mdanderson.org